CLINICAL TRIAL: NCT07226102
Title: An E-Health Intervention for Fear of Progression in Women With Gynecologic or Breast Cancer
Brief Title: Virtual Mental Health Intervention to Address Fear of Progression for Women With High Risk or Stage III-IV Gynecologic or Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 24425; NCI-2025-07274 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24425 (Other: CITY OF Hope Medical Center); P30CA033572 (NIH); R21CA293326 (NIH)
Record Dates: First submitted 2025-10-16; First posted 2025-11-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Endometrial Carcinoma; Endometrial Endometrioid Adenocarcinoma; Female Reproductive System Neoplasm; Stage II Ovarian Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Vaginal Cancer AJCC v8; Stage III Vulvar Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Vaginal Cancer AJCC v8; Stage IV Vulvar Cancer AJCC v8; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms; Genital Neoplasms, Female; Ovarian Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Triple Negative Breast Neoplasms | interventions — Behavior Therapy; Early Intervention, Educational; Educational Status; Methods; Interviews as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Following completion of baseline questionnaires and the intake call, the clinical research assistant will be informed of the group assignment. The study team is blinded to assignment until this point. The study participants will be blinded to group assignment (single-blind).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Fear of progression intervention) (Experimental): Patients receive access to the Day by Day platform that includes patient partner videos, testimonials, handouts and a community forum. Patients may optionally utilize these resources for 6 weeks. Patients attend online group sessions, over 60 minutes, for every other week for 3 sessions and complete online educational sessions on values clarification, managing worry and unhelpful thoughts, and skills practices to promote healthy coping on alternate weeks for 3 sessions. Patients complete a check in call, for 15-20 minutes, at week 3-4. Patients are asked to practice the skills including attention training, mindfulness, worry postponement, guided imagery and other practices from the intervention for 10-12 minutes, at least 6 days per week for and track their practice on the Day to Day platform for 6 weeks. Patients may be loaned a tablet if needed for 6 weeks.
  Interventions: Behavioral: Behavioral Intervention; Other: Educational Intervention; Other: Internet-Based Intervention; Other: Interview; Other: Survey Administration; Other: Virtual Technology Intervention
- Arm II (Educational intervention) (Active Comparator): Patients receive access to the Empower Hope platform. Patients attend online group sessions, over 60 minutes, for every other week for 3 sessions and complete online educational sessions on clinical trial participation, identifying reliable online information, healthy living on nutrition and activity/exercise and coping with fatigue on alternate weeks for 3 sessions. Patients complete a check in call, for 15-20 minutes, at week 3-4. Patients may be loaned a tablet if needed for 6 weeks.
  Interventions: Behavioral: Behavioral Intervention; Other: Educational Intervention; Other: Internet-Based Intervention; Other: Interview; Other: Survey Administration; Other: Virtual Technology Intervention

INTERVENTIONS:
Behavioral: Behavioral Intervention — Attend online group sessions
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm I (Fear of progression intervention)
Behavioral: Behavioral Intervention — Complete online educational sessions
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm I (Fear of progression intervention)
Behavioral: Behavioral Intervention — Complete check in call
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
Behavioral: Behavioral Intervention — Complete daily skills practice
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm I (Fear of progression intervention)
Other: Educational Intervention — Receive access to patient partner videos, testimonials, handouts and a community forum
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm I (Fear of progression intervention)
Other: Educational Intervention — Attend online group sessions
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm II (Educational intervention)
Other: Educational Intervention — Complete online education sessions
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm II (Educational intervention)
Other: Internet-Based Intervention — Receive access to Day to Day platform
  Arms: Arm I (Fear of progression intervention)
Other: Internet-Based Intervention — Receive access to the Empower Hope platform
  Arms: Arm II (Educational intervention)
Other: Interview — Ancillary studies
Other: Survey Administration — Ancillary studies
Other: Virtual Technology Intervention — Receive a tablet
  Other Names: Virtual Reality Intervention; Virtual Technology

SUMMARY:
This clinical trial tests feasibility, acceptability and how well a virtual mental health intervention, compared to enhanced usual care consisting of an educational intervention, works to address fear of progression for women with high risk or stage III-IV gynecologic or breast cancer. Worrying about cancer coming back or progression is natural for cancer patients. Many cancer patients face stress and uncertainty as they live longer and attend regular check-ups. A supportive program can help to develop skills to feel calmer and more resilient during uncertain times and better manage feelings of fear. The virtual mental health intervention may be a feasible, acceptable and effective may to address fear of progression for women with high risk or stage III-IV gynecologic or breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility and acceptability of a blended e-health intervention to manage fear of progression (FOP) in patients with stage III or IV gynecologic (GYN) or breast cancer.

SECONDARY OBJECTIVE:

I. To determine the effects of the intervention on reducing fear of cancer progression (FOP) (primary outcome) and improving secondary outcomes of distress, anxiety, metacognitions, and mindfulness.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive access to the Day by Day platform that includes patient partner videos, testimonials, handouts and a community forum. Patients may optionally utilize these resources for 6 weeks. Patients attend online group sessions, over 60 minutes, for every other week for 3 sessions and complete online educational sessions on values clarification, managing worry and unhelpful thoughts, and skills practices to promote healthy coping on alternate weeks for 3 sessions. Patients complete a check in call, for 15-20 minutes, at week 3-4. Patients are asked to practice the skills including attention training, mindfulness, worry postponement, guided imagery and other practices from the intervention for 10-12 minutes, at least 6 days per week for and track their practice on the Day to Day platform for 6 weeks. Patients may be loaned a tablet if needed for 6 weeks.

ARM II: Patients receive access to the Empower Hope platform. Patients attend online group sessions, over 60 minutes, for every other week for 3 sessions and complete online educational sessions on clinical trial participation, identifying reliable online information, healthy living on nutrition and activity/exercise and coping with fatigue on alternate weeks for 3 sessions. Patients complete a check in call, for 15-20 minutes, at week 3-4. Patients may be loaned a tablet if needed for 6 weeks.

After completion of study intervention, patients are followed up at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women with stage III or IV GYN (ovarian, endometrial, cervical, vulvar/vaginal) or breast cancer who are at least 2 months from initial diagnosis
* Women with high-risk disease e.g., carcinosarcoma; ovarian cancer stage II or grade III histology; endometrioid endometrial cancer stage II or III; grade III with LVI or deep invasion; serous, clear cell or undifferentiated histologies; triple negative breast cancer
* Score ≥ 34 on the Fear of Progression Short-Form, indicating dysfunctional levels
* Age 18 or older; able to read and understand English
* Patients in remission or with progressive disease

Exclusion Criteria:

* Enrolled in hospice
* Major depression as assessed by patient health questionnaire (PHQ)-9
* Non-English speaking
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-07-16 (Estimated); Primary Completion 2026-07-16 (Estimated); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Fear of cancer progression (FOP-SF) | Baseline, 6 weeks, up to 12 weeks
  FOP-SF consists of 12 items pertaining to 4 subscales: affective reactions; partnership/family; occupation; loss of autonomy. Scores range from 12-60; higher levels indicate greater FOP; a cut-off of 34 and above indicates dysfunctional FOP levels. The FOP-SF has been validated in a large sample of breast and mixed cancer patients (a=.87) patients who completed a rehabilitation program (a=.90). The correlation between the long and short form of the questionnaires is r=0.92. Validity has been demonstrated by correlation with HADS anxiety (r=.65 to .71), GAD anxiety (r=.57) and depression (r=.49). In a descriptive FOP study in 135 English-speaking cancer survivors, the FOP-SF showed high internal consistency (a=0.88) and was correlated with similar constructs: Intrusions (r=.72), metacognitive beliefs (r=0.62); death anxiety (r=0.67) (Curran et al., 2020).

SECONDARY OUTCOMES:
Cancer-related distress - Impact of Event Scale-R (IES-R) | Baseline, 6 weeks, Up to 12 weeks
  The IES-R measures cancer-related distress. It consists of 22-likert-scale items representing 3 subscales: Intrusion; Avoidance; and Hyperarousal. Items are scored on a 0-4 response format. Total scores range from 0-88. A score of 24 or greater indicates clinical levels of distress. It demonstrates good internal consistency; a=.79-.92. The IES has been used in several studies with cancer patients. It has been found to be sensitive to change in these interventions (Butow et al. 2017).
Anxiety - PROMIS - Anxiety 8-a | Baseline, 6 weeks, Up to 12 weeks
  This measures fear, worry, hyperarousal, and related somatic symptoms (Cella et al., 2010). It consists of 8 items scored on a 0-5 response format. Scores are standardized to continuous T scores with a mean of 50 and SD of 10; higher scores reflect higher distress. PROMIS T score thresholds for anxiety are less than 55 normal; 55-64 mild; 65-74 moderate; greater than or equal to 75 severe. Validity was established in a large sample of patients with chronic illnesses, including cancer. Construct validity was demonstrated using the anxiety scale from the MASQ as the convergent measure (r=.80) and the CES-D as the divergent measure (r=.75).
Metacognitive Beliefs - Metacognitions questionnaire (MCQ-18) | Baseline, 6 weeks, Up to 12 weeks
  The MCQ assesses different beliefs about worry. We will use 18 items from three subscales of the parent MCQ-30 questionnaire a) positive beliefs about worry; b) negative beliefs about worry; and c) need to control thoughts. Items are scored on a 1-4 Likert scale. Subscale scores range from 6-24. Higher scores indicate more dysfunctional metacognitions. Internal consistency was a=.93 for the total score and ranged from .72-.93 for the subscale scores. It has been validated in cancer patients showing good convergent validit7 (Cook et al., 2014). Internal consistency of the subscales ranged from .73-.89 (pre-treatment) and .79-.91 (post-treatment).
Mindfulness - Five Facet Mindfulness Questionnaire (FFMQ-15) | Baseline, 6 weeks, Up to 12 weeks
  FFMQ-15 assesses 5 facets of mindfulness: Observing, Describing, Acting with awareness, non-reactivity to inner experience, and non-judging of inner experience. Items are rated on a 5-point Likert scale ranging from 1-5 scale (never/ rarely to very often). Three items comprise each subscale. Subscale scores range from 3-15. Higher scores indicate greater mindfulness skills engagement. The measure is sensitive to change over the course of mindfulness-based cognitive therapy (Chambers et al., 2017). For scoring, the Observing subscale score is excluded based on psychometric testing data from previous research. The total FFMQ score is calculated by summing the 4 subscale scores. For the subscales, internal consistency is adequate (a=.66-.83) (Baer et al., 2006). The FFMQ has been used in studies of advanced cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Reb, Principal Investigator — City of Hope Medical Center
Locations (12):
- United States (12):
  - City of Hope at Arcadia, Arcadia, California
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope at Long Beach Worsham, Long Beach, California
  - City of Hope at Long Beach Elm, Long Beach, California
  - City of Hope Mission Hills, Mission Hills, California
  - City of Hope - Santa Clarita, Santa Clarita, California
  - City of Hope at Simi Valley, Simi Valley, California
  - City of Hope at Thousand Oaks, Thousand Oaks, California
  - City of Hope South Bay, Torrance, California
  - City of Hope Upland, Upland, California